CLINICAL TRIAL: NCT00722943
Title: Neuroendocrine Mechanisms of Developmental Massage Therapy (DMT) in Preterm Infants: Clinical Study
Acronym: DMT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 28032
Record Dates: First submitted 2008-07-24; First posted 2008-07-28 (Estimated); Last update posted 2013-02-08 (Estimated); Status verified 2013-02

CONDITIONS: Premature Birth of Newborn
Keywords: infant; premature; message; therapy; NICU; neonatal intensive care unit; cortisol level; stress; postnatal; weight gain; DMT; Development Message Therapy; growth
MeSH Terms: conditions — Premature Birth; Weight Gain

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DMT group (Active Comparator): These infants will receive tactile stimulation and developmental massage by a licensed therapist. This intervention will be done behind a screen in order to blind the therapy to NICU staff and parents.
  Interventions: Other: Developmental Massage Therapy
- SHAM control (Placebo Comparator): These infants will have no tactile stimulation or developmental massage done. The therapist will stand behind a screen but will not touch the infant. The screen will blind the NICU staff and parents to the study arm.
  Interventions: Other: no intervention

INTERVENTIONS:
Other: Developmental Massage Therapy — Tactile stimulation and massage will be done by a licensed therapist
  Arms: DMT group
Other: no intervention — The infant will not be touched by the therapist.
  Arms: SHAM control

SUMMARY:
The purpose of this study is to see if daily massage therapy will help premature infants respond to stress better, as well as improve their growth and neurobehavioral development.

DETAILED DESCRIPTION:
Optimal postnatal growth and development is essential for the survival and long-term health of infants born premature, however, growth and developmental delays are common. Many factors contribute to poor postnatal growth and development including immature organ systems, stress due to illness and even routine care in the neonatal intensive care unit environment. Massage therapy is associated with decreased cortisol levels during stress in a variety of populations including premature infants. Massage has also been reported to improve postnatal weight gain in premature infants. Concerns about methodological quality, however, weaken the credibility of previous studies and prevent the integration of massage therapy into conventional medical practice. Therefore, we plan to study the interrelationship of the ANS and HPA axis in preterm infants to assess how developmental massage therapy (DMT) modulates physiologic stability and promotes postnatal growth by the following specific aims:

SPECIFIC AIM 1: We will determine ANS balance, measured by heart period variability, before, during, and after DMT.

SPECIFIC AIM 2: We will compare the relationships between ANS balance and HPA response before and after DMT.

SPECIFIC AIM 3: We will evaluate somatotrophic response in premature infants who receive DMT.

Infants will be stratified by gender and randomized to receive developmental massage therapy or SHAM control.

This study will also allow for post-discharge assessment of development. Infants will return to the hospital at term, 3months and 6 months for multiple measurements and developmental testing.

ELIGIBILITY:
Inclusion Criteria:

* Premature infants born between 29 4/7 and 32 3/7 weeks gestation by physical exam at birth, and with birth weight, length and head circumference between the 5th and 95th percentiles for gestational age.

Exclusion Criteria:

* Intrauterine growth less than the 5th or greater than the 95th percentiles for gestational age, congenital anomalies, complex cardiac defects, severe CNS injury, hypothyroidism, inborn errors of metabolism, or inability to establish full enteral feeds by day of life 14.

Max Age: 14 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 46 (Actual)
Dates: Start 2008-07; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Growth | Weekly

SECONDARY OUTCOMES:
Salivary cortisol levels | Daily for first week; Weekly thereafter
Neurobehavioral Assessment | Weekly, Term, 3 months, 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Laurie J Moyer-Mileur, PhD, Principal Investigator — University of Utah
Locations (3):
- United States (3):
  - Intermountain Medical Center, Murray, Utah
  - St. Mark's Hospital, Salt Lake City, Utah
  - University of Utah, Salt Lake City, Utah

REFERENCES:
- [Derived] Moyer-Mileur LJ, Haley S, Slater H, Beachy J, Smith SL. Massage improves growth quality by decreasing body fat deposition in male preterm infants. J Pediatr. 2013 Mar;162(3):490-5. doi: 10.1016/j.jpeds.2012.08.033. Epub 2012 Oct 11. PMID 23062248